CLINICAL TRIAL: NCT07407803
Title: Randomized, Double-Blind, Parallel-Controlled, Multicenter Phase III Clinical Trial Evaluating the Efficacy and Safety of TQ-B3234 Capsules Versus Placebo in Patients With Symptomatic, Non-Surgical Type 1 Neurofibromatosis-Associated Plexiform Neurofibromas
Brief Title: Evaluation of TQ-B3234 Capsules in Patients With Symptomatic, Non-Surgical Type 1 Neurofibromatosis-Associated Plexiform Neurofibromas
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQ-B3234-III-01
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Plexiform Neurofibroma
MeSH Terms: conditions — Neurofibroma, Plexiform

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-B3234 capsules (Experimental): TQ-B3234 capsules: 50 mg once daily, one cycle every 4 weeks (28 days)
  Interventions: Drug: TQ-B3234 capsules
- TQ-B3234 placebo (Placebo Comparator): TQ-B3234 placebo: 0 mg once daily, one cycle every 4 weeks (28 days)
  Interventions: Drug: TQ-B3234 placebo

INTERVENTIONS:
Drug: TQ-B3234 capsules — TQ-B3234 is an antitumor molecular targeted drug, a selective mitogen-activated protein kinase 1 and 2 (MEK1/2) inhibitor. It primarily inhibits the mitogen-activated protein kinase (MEK) protein (an upstream regulator of the extracellular signal-regulated kinase (ERK) pathway), thereby affecting the mitogen-activated protein kinase (MAPK) pathway and suppressing cell proliferation. MEK inhibitors are recognized to play a significant role in the pathogenesis of plexiform neurofibromas associated with neurofibromatosis type 1.
  Arms: TQ-B3234 capsules
Drug: TQ-B3234 placebo — TQ-B3234 placebo without drug substance.
  Arms: TQ-B3234 placebo

SUMMARY:
This study aims to demonstrate that in subjects with symptomatic, inoperable plexiform neurofibromas associated with neurofibromatosis type 1, TQ-B3234 capsules significantly improve the objective response rate at Week 24 compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* The subject voluntarily joins this study, signs the informed consent form, and demonstrates good compliance.
* Age ≥18 years (calculated from the date of signing the informed consent form).
* Diagnosis of symptomatic, non-resectable neurofibromatosis type 1 (NF1)-associated plexiform neurofibroma (PN) requiring systemic therapy per investigator judgment.
* At least one measurable lesion with a dimension ≥3 cm.
* There should be no significant changes in the use of chronic neuropathic pain medications within 28 days prior to study enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Laboratory tests meet the protocol criteria.
* Women of childbearing potential must agree to use effective contraception during the study and for 6 months after study completion. A negative serum pregnancy test must be documented within 7 days prior to study enrollment. Men must agree to use effective contraception during the study and for 6 months after study completion.

Exclusion Criteria:

* Confirmed or suspected malignant glioma or malignant peripheral nerve sheath tumor (MPNST) (excluding low-grade glioma, optic nerve glioma not requiring systemic therapy or radiotherapy); histological confirmation may be required.
* History of or concurrent other malignancies within 5 years prior to first dosing.
* Multiple factors affecting oral drug absorption (e.g., dysphagia, chronic diarrhea, intestinal obstruction, major bowel resection).
* Adverse reactions from prior anti-tumor therapy not recovered to NCI CTCAE v6.0 grade ≤1, except grade 2 alopecia, grade 2 peripheral neuropathy, grade 2 anemia, non-clinically significant and asymptomatic laboratory abnormalities, and hypothyroidism stabilized by hormone replacement therapy.
* Major surgery, significant traumatic injury, or planned major surgery during the study within 4 weeks prior to first dosing; or presence of long-term non-healed wounds or fractures.
* History of arterial/venous thrombotic events (e.g., cerebrovascular accident including transient ischemic attack (TIA), deep vein thrombosis, pulmonary embolism) or other severe thromboembolic events within 6 months prior to first dosing.
* Active viral hepatitis with poor control.
* Active syphilis requiring treatment.
* Active tuberculosis, idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonia, radiation pneumonitis requiring treatment, or clinically symptomatic active pneumonia.
* History of substance abuse that cannot be controlled or presence of psychiatric disorders.
* Planned or prior allogeneic bone marrow or solid organ transplantation.
* History of hepatic encephalopathy.
* History of or current retinal vein occlusion (RVO), retinal pigment epithelial detachment (RPED), central serous retinopathy (CSR), glaucoma, or other significant ocular abnormalities (e.g., intraocular pressure >21mmHg).
* Inability to undergo MRI and/or presence of MRI contraindications.
* Major cardiovascular disease.
* Active or uncontrolled severe infection.
* Renal failure requiring hemodialysis or peritoneal dialysis.
* History of immunodeficiency, including HIV-positive or other acquired/congenital immunodeficiency diseases.
* History of epilepsy.
* Tumor-related symptoms and treatment.
* Known hypersensitivity to study drug excipients.
* Participation in and use of other PN clinical trial drugs within 4 weeks prior to first dosing.
* Pregnant or lactating participants.
* Any other condition that, in the investigator's judgment, poses a serious risk to participant safety or interferes with study completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
IRC-Assessed Objective Response Rate (ORR) | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Percentage of subjects achieving complete response (CR) or partial response (PR) as assessed by independent review committee (IRC) per REiNS criteria at the end of Cycle 24.

SECONDARY OUTCOMES:
Investigator-Assessed ORR | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Percentage of subjects achieving complete response (CR) or partial response (PR) as assessed by investigators per REiNS criteria.
IRC/Investigator-Assessed DOR | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Duration of response (DOR), defined as the time from first documented confirmed objective response to disease progression or death from any cause (whichever occurs first), as determined by IRC/investigators per REiNS criteria.
IRC/Investigator-Assessed disease control rate (DCR) | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Percentage of subjects achieving complete response (CR), partial response (PR), or stable disease (SD) as determined by IRC/investigators per REiNS criteria.
IRC/Investigator-Assessed progression-free survival (PFS ) | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Time from randomization to first disease progression or death from any cause (whichever occurs first), as determined by IRC/investigators per REiNS criteria.
IRC/Investigator-Assessed TTP | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Time from randomization to first disease progression (TTP), as assessed by IRC/investigators per REiNS criteria.
IRC/Investigator-Assessed time to response (TTR) | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Time from randomization to first objective response, as determined by IRC/investigators per REiNS criteria.
Tumor response in subject | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Difference in the best percentage change from baseline in target PN volume between groups, as assessed by IRC/investigators.
Number of subjects with incidence and severity of adverse events (AEs) | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Incidence and severity of adverse events from subject enrollment to the end of cycle 24.
Patient-reported outcomes | From subject enrollment to the end of cycle 24 (each cycle is 28 days)
  Patient self-assessment results from subject enrollment to the end of cycle 24.
Peak concentration (Cmax) | 2 hours after administration
  Maximum plasma drug concentration
Plasma concentration at steady state (Ctrough, SS) | Cycle 1 day 28: pre-dose, Cycle 2 day 28 pre-dose, Cycle 3 day 28: pre-dose, Cycle 6 day 28: pre-dose. (each cycle is 28 days)
  The pre-dose concentration observed when the drug has reached steady state with repeated dosing, indicating baseline exposure and accumulation.
Effects on pain score in subjects | From subject enrollment to the end of the 24th cycle (each cycle is 28 days)
  Questionnaire: Numerical Rating Scale-11 (NRS-11); The line segments below all have numbers from 0 to 10, where 0 means no pain and 10 is the worst pain you can imagine.
Effects on pain interference index in subjects | From subject enrollment to the end of the 24th cycle (each cycle is 28 days)
  Questionnaire: pain interference index; Please answer each one by circling a number from 0 to 6, where 0 means none at all and 6 means completely
Effects on subjects' general quality of life | From subject enrollment to the end of the 24th cycle (each cycle is 28 days)
  Questionnaire: Functional Assessment of Cancer Therapy - General (FACT-G); the scores from all items across its four domains are summed to obtain a total score, which ranges from 0 to 108 points.
Effects on subjects; disease-specific quality of life | From subject enrollment to the end of the 24th cycle (each cycle is 28 days)
  Questionnaire: PedsQL NF1 Module; It includes an Adult version (>25 years) and a Young Adult version (18-25 years), with 104 items, respectively.

CONTACTS AND LOCATIONS:
Locations (28):
- China (28):
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality
  - Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking University Third Hospital, Beijing, Beijing Municipality
  - The Southwest Hospital of Amu, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujan Medical University, Fuzhou, Fujian
  - Gansu Provincial Cancer Hospital, Lanzhou, Gansu
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Dermatology Hospital of Southern Medical University (Guangdong Provincial Dermatology Hospital / Guangdong Center for the Prevention and Control of Sexually Transmitted Diseases and Leprosy, Guangzhou, Guangdong
  - Guangxi Medical University Cancer Hospital （ Guangxi Cancer InstituteGuangxi Cancer Hospital & Medical University Oncology School & Cancer Center）, Nanning, Guangxi
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The second hospital of Hebei medical university, Shijiazhuang, Hebei
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - The First Affiliated Hospital Of Zhengzhou University, Zhengzhou, Henan
  - Renmin Hospital of Wuhan University(Hubei General Hospital), Wuhan, Hubei
  - Hunan Children's Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Xijing hospital, Xi'an, Shaanxi
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shanghai Ninth People's Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Sichuan Academy of Medical Science&Sichuan Provincial People' Hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital Of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Provincial People'S Hospital, Hangzhou, Zhejiang